CLINICAL TRIAL: NCT06698718
Title: Application of CIELab Spectrophotometry to Analyze Gingival Color: a New Perspective for Evaluating the Effectiveness of Periodontal Basic Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-0935
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Periodontitis
Keywords: periodontitis; Periodontal basic treatment; Spectrophotometer colorimeter
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Procedure: Periodontal basic treatment

INTERVENTIONS:
Procedure: Periodontal basic treatment — Accept periodontal basic treatment

SUMMARY:
Objective: This study aims to explore the correlation between gingival color and clinical indicators and inflammatory factors in patients with periodontitis.

Method: This study aims to include 30 periodontitis patients who visited the Periodontology Department of the Second Affiliated Hospital of Zhejiang University School of Medicine from October 2024 to November 2024. The study adopted a self controlled before and after design. All subjects received periodontal basic treatment. Record the age, gender, ethnicity, skin color, and gingival biotype of the subjects. Before treatment, 6 weeks after treatment, and 12 weeks after treatment, check and record the blood routine, high-sensitivity C-reactive protein (Hs CRP), and interleukin-6 (IL-6) of all subjects. Use a moisture absorbing paper tip to collect the gingival crevicular fluid of the subjects, and further detect the levels of interleukin-17 (IL-17) and tumor necrosis factor alpha (TNF - α) in the gingival crevicular fluid samples, and record the periodontal table. Check and record the CIE indicators L *, a *, b *, probing depth (PD), gingival bleeding index (SBI), and clinical attachment loss (CAL) in the keratinized gingival area of all subjects before and after treatment at 2, 6, and 12 weeks. Analyze and compare the changes in each group's data before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of Han ethnicity, aged between 18 and 65 years old, diagnosed with periodontitis
2. I haven't received any periodontal basic treatment, including scaling, scraping, flap surgery, etc., for the past six months
3. The anterior teeth area has not undergone periodontal surgery or coronal restoration within six months
4. The patient has clear thinking, unobstructed communication, and high compliance

Exclusion Criteria:

1. Cardiac function levels III and IV
2. Blood pressure>180/110 mmHG
3. Pregnant women, women in pregnancy or lactation
4. Those who are currently taking anticoagulant drugs, calcium channel blockers, immunosuppressants, angiotensin and other medications, receiving bisphosphonates treatment, or have a history of antibacterial treatment within 3 months
5. Uncontrolled and stable patients with systemic diseases, such as progressive liver diseases, infectious diseases, renal failure, rheumatoid diseases, blood system diseases, osteoporosis, AIDS, mental diseases and diabetes, etc
6. Patients with malignant tumors or undergoing radiotherapy, chemotherapy, and targeted drug therapy
7. Patients with pacemakers who cannot undergo ultrasound therapy
8. Smoking or quitting smoking for less than 5 years
9. Individuals with abnormalities such as pigment deposition and keratinized beads in the front teeth and gums

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
CIE indicators L *, a *, b for keratinized gingival area in the anterior teeth region* | 12 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China